CLINICAL TRIAL: NCT00192933
Title: Evaluation of the Quality of the NovoSeven (rFVIIa) Tratment Practice at Rigshospitalet, Copenhagen University Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Other Study IDs: 2004-41-3996
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2006-10-19 (Estimated); Status verified 2005-09

CONDITIONS: Hemorrhage; Shock
MeSH Terms: conditions — Hemorrhage; Shock

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Procedure: NovoSeven treatment according to guideline

SUMMARY:
The purpose is to evaluate and improve NovoSeven treatment practice done according to our guidelines

ELIGIBILITY:
Inclusion Criteria:

* Indication for NovoSeven treatment according to our guideline

Exclusion Criteria:

-

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-01; Study Completion 2010-12

CONTACTS AND LOCATIONS:
Overall Officials: Pär Johansson, MD, MPA, Study Chair — Blood Bank, Rigshospitalet, Copenhagen University Hospital
Locations (1):
- Rigshospitalet, Copenhagen University Hospital, Copenhagen, Denmark